CLINICAL TRIAL: NCT00353704
Title: Analgetic and Anxiolytic Effect of Preoperative Pregabalin in Patients Undergoing Surgery of the Vertebral Columna
Brief Title: Analgetic and Anxiolytic Effect of Preoperative Pregabalin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Ulrich Johannes Spreng, Asker and Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-003229-20
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Intervertebral Disk Displacement; Disk Prolapse
Keywords: Intervertebral disk displacement; disk prolapse; pregabalin
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Pregabalin; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Pregabalin (Active Comparator): 150 mg Pregabalin per orally about one hour before surgery
  Interventions: Drug: pregabalin; Drug: morphine
- Placebo (Placebo Comparator): One capsule of saccharose (placebo) was administered orally about one hour before surgery.
  Interventions: Drug: Placebo; Drug: morphine

INTERVENTIONS:
Drug: pregabalin — capsule 150 mg x 1 per orally one hour before surgery
  Arms: Pregabalin
Drug: Placebo — One capsule of saccharose (placebo) was administered about one hour before surgery
  Arms: Placebo
Drug: morphine — All patients were equipped with a PCA (patient controlled analgesia) for 24 hours after surgery. The sum of morphine used was registered (milligram).

SUMMARY:
The purpose of this study is to determine whether the use of oral pregabalin 150 mg as premedication reduces the amount and degree of postoperative pain.

Furthermore the purpose of this study is to determine whether the use of oral pregabalin 150 mg as premedication reduces anxiety prior to anaesthesia in these patients.

DETAILED DESCRIPTION:
The mechanism of development of postoperative pain is complex. Central and peripheral sensitization are playing an important role and this can lead to postoperative hypersensitization. Several studies have shown, that gabapentin can be effective to reduce sensitization and postoperative pain. Pregabalin (S-aminomethyl-5-methylhexaninacid) is a further development of gabapentin. Pregabalin has a fewer side-effects compared with gabapentin.

The purpose of this study is to compare the analgetic and anxiolytic effect of pregabalin and placebo used as premedication.

The hypothesis is that a single-dose pregabalin (150 mg postoperatively (p.o.)) gives significant better anxiolysis and analgesia than placebo.

The study is including patients undergoing surgery of the vertebral columna.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of disc prolapse
* Age 18+
* ASA (American Association in Anesthesiology) I-III
* written consent

Exclusion Criteria:

* Age < 18
* ASA > III
* liver failure
* renal failure
* allergic reaction against gabapentin and/or pregabalin
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-11; Primary Completion 2009-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich J Spreng, Dr. med., Principal Investigator — Asker and Baerum Hospital, Norway; Vegard Dahl, Dr. med., Study Director — Asker and Baerum Hospital, Norway
Locations (1):
- Asker and Baerum Hospital, Rud, Norway

REFERENCES:
- [Background] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Background] Menigaux C, Adam F, Guignard B, Sessler DI, Chauvin M. Preoperative gabapentin decreases anxiety and improves early functional recovery from knee surgery. Anesth Analg. 2005 May;100(5):1394-1399. doi: 10.1213/01.ANE.0000152010.74739.B8. PMID 15845693
- [Background] Dirks J, Fredensborg BB, Christensen D, Fomsgaard JS, Flyger H, Dahl JB. A randomized study of the effects of single-dose gabapentin versus placebo on postoperative pain and morphine consumption after mastectomy. Anesthesiology. 2002 Sep;97(3):560-4. doi: 10.1097/00000542-200209000-00007. PMID 12218520
- [Derived] Spreng UJ, Dahl V, Raeder J. Effect of a single dose of pregabalin on post-operative pain and pre-operative anxiety in patients undergoing discectomy. Acta Anaesthesiol Scand. 2011 May;55(5):571-6. doi: 10.1111/j.1399-6576.2011.02410.x. Epub 2011 Mar 8. PMID 21385158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period november 2005 until june 2008
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 25 | 25
Completed | 22 | 24
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 43 (8) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Norway | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean VAS Pain (Visual Analogue Scale)at Rest (0-100 mm)
Description: The visual analogue scale (VAS) was used for registration of the pain intensity at rest. The score ranges from 0-100, where 0 means no pain and 100 means maximal pain. Higher values represent a worse outcome.
Time Frame: 120 minutes after surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 24
Units on a scale | 11.7 (9.6) | 22.5 (14.4)

2. Secondary Outcome: Morphine (Opioid) Consumption Cumulated
Description: Patients were equipped with a morphine PCA (patient controlled analgesia) for 24 hours after surgery. So they could administrate morphine intravenously by pressing a button. The sum of morphine was registered as " cumulated opioid consumption (milligram)
Time Frame: 240 minutes
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 24
mg | 7.3 (6.3) | 16.0 (13.2)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes